CLINICAL TRIAL: NCT05543954
Title: A Pilot Study of 68Ga-FAPI-RGD PET/CT Imaging in the Lung Cancer Patients
Brief Title: 68Ga-FAPI-RGD PET/CT Imaging in the Lung Cancer Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-NM-FR
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Fluorodeoxyglucose F18; 68Ga-FAPI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 68Ga-FAPI-RGD and 18F-FDG PET/ CT scan (Experimental): Within 2 week, each patient underwent PET/CT scan after intravenous administration of 68Ga-FAPI-RGD and 18F-FDG, respectively.
  Interventions: Drug: 68Ga-FAPI-RGD; Drug: 18F-FDG
- 68Ga-FAPI-RGD and 68Ga-FAPI PET/ CT scan (Experimental): Within 2 week, each patient underwent PET/CT scan after intravenous administration of 68Ga-FAPI-RGD and 68Ga-FAPI, respectively.
  Interventions: Drug: 68Ga-FAPI-RGD; Drug: 68Ga-FAPI
- 68Ga-FAPI-RGD and 68Ga-RGD PET/ CT scan (Experimental): Within 2 week, each patient underwent PET/CT scan after intravenous administration of 68Ga-FAPI-RGD and 68Ga-RGD, respectively.
  Interventions: Drug: 68Ga-FAPI-RGD; Drug: 68Ga-RGD

INTERVENTIONS:
Drug: 68Ga-FAPI-RGD — Intravenous injection of 68Ga-FAPI-RGD with a dosage of approximately 1.8-2.2 MBq (0.05-0.06 mCi)/kg.
  Other Names: 68Ga-FAPI-RGD injection
Drug: 18F-FDG — Intravenous injection of 18F-FDG with a dosage of approximately 3.7-5.55 MBq (0.1-0.15 mCi)/kg.
  Other Names: 18F-FDG injection
  Arms: 68Ga-FAPI-RGD and 18F-FDG PET/ CT scan
Drug: 68Ga-FAPI — Intravenous injection of 68Ga-FAPI with a dosage of approximately 1.8-2.2 MBq (0.05-0.06 mCi)/kg.
  Other Names: 68Ga-FAPI injection
  Arms: 68Ga-FAPI-RGD and 68Ga-FAPI PET/ CT scan
Drug: 68Ga-RGD — Intravenous injection of 68Ga-RGD with a dosage of approximately 1.8-2.2 MBq (0.05-0.06 mCi)/kg.
  Other Names: 68Ga-RGD injection
  Arms: 68Ga-FAPI-RGD and 68Ga-RGD PET/ CT scan

SUMMARY:
Based on the high expression of specific receptors on the surface of diseased tissues and neovascularization, noninvasive targeted molecular imaging can be used to visualize lesions in vitro by combining specific ligands labeled with short half-life isotopes. Lung cancer tissues express fibroblast activating protein FAP, and also have high expression of integrin αVβ3 receptor on the surface of blood vessels. In this study, a novel dual-target imaging agent 68Ga-FAPI-RGD was used for PET/CT imaging of lung cancer.

DETAILED DESCRIPTION:
Conventional 18F-FDG PET/CT has important diagnostic value in cell metabolism level, early metastasis, judging malignant potential and prognosis of tumors. It has been routinely used for staging and restaging of most tumors, but there are still some tumors with low uptake of 18F-FDG PET/CT. Moreover, 18F-FDG cannot distinguish between tumors and inflammatory diseases, such as tuberculosis and granuloma. Receptor imaging with a single target also has some limitations in clinical application. For example, not all diseased cells express a large amount of single receptor on the surface, which greatly affects the judgment of the nature of the lesion. The dual-target molecular imaging based on FAP expressed in the lesion site and integrin αvβ3 receptor highly expressed on the surface of the lesion neovascularization will overcome the above limitations and make full use of the advantages of the dual-target molecular imaging, which will greatly assist the diagnosis of malignant tumors such as lung cancer. In this study, a novel dual-target imaging agent 68Ga-FAPI-RGD was used for PET/CT imaging of lung cancer, compared with conventional 18F-FDG, or single target imaging agent 68Ga-RGD or 68Ga-FAPI PET/CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed or suspected lung cancer;
* 68Ga-FAPI-RGD and 18F-FDG(or 68Ga-FAPI or 68Ga-RGD) PET/CT within 2 week;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance1 | through study completion, an average of 1 year
  comparing the SUV and number of lung cancer or metastasis detected by 68Ga-FAPI-RGD and 18F-FDG PET/CT
Diagnostic performance2 | through study completion, an average of 1 year
  comparing the SUV and number of lung cancer or metastasis detected by 68Ga-FAPI-RGD and 68Ga-FAPI PET/CT
Diagnostic performance3 | through study completion, an average of 1 year
  comparing the SUV and number of lung cancer or metastasis detected by 68Ga-FAPI-RGD and 68Ga-RGD PET/CT

SECONDARY OUTCOMES:
The dosimetry of 68Ga-FAPI-RGD | through study completion, an average of 1 year
  Measure the distribution of 68Ga-FAPI-RGD in 6-8 lung cancer patients by 3-hour dynamic PET/CT acquisition by dosimetry software
68Ga-FAPI-RGD uptake at different time points | through study completion, an average of 1 year
  The SUV uptake of tumors and metastases in patients with lung cancer was measured at 1, 2, and 3 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD,PHD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China